CLINICAL TRIAL: NCT00781924
Title: Interventional Sonography Guided by Image Fusion
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Caroline Ewertsen, Rigshospitalet
Other Study IDs: HD-2007-0066
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2009-08

CONDITIONS: Focal Liver Lesions; Focal Lesions in the Abdomen
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- biopsy
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — ultrasound guided biopsy of tumors.

SUMMARY:
The purpose of this study is to register the precision of image fusion between live sonography and CT, MRI or PET/CT of liver lesions and other focal lesions in the abdomen. To test whether it will be possible to biopsy guided by image fusion.

ELIGIBILITY:
Inclusion Criteria:

* Focal liver lesion seen on CT, MRI or PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with focal liver lesions where biopsy is needed or the lesion has to be verified by sonography
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Verification of the tumor by sonography | baseline only

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Ewertsen C, Henriksen BM, Hansen CP, Knigge U. Synchronous gastric neuroendocrine carcinoma and hepatocellular carcinoma: a case report. BMJ Case Rep. 2009;2009:bcr03.2009.1667. doi: 10.1136/bcr.03.2009.1667. Epub 2009 Sep 15. PMID 21918674